CLINICAL TRIAL: NCT02420756
Title: Imaging Dementia-Evidence for Amyloid Scanning (IDEAS) Study: A Coverage With Evidence Development Longitudinal Cohort Study
Brief Title: Imaging Dementia-Evidence for Amyloid Scanning (IDEAS) Study
Acronym: IDEAS
Status: Completed | Type: Observational
Sponsor: American College of Radiology (Other)
Collaborators: Alzheimer's Association (Other); American College of Radiology Imaging Network (Network)
Responsible Party: Sponsor
Other Study IDs: IDEAS Study
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Alzheimer's Disease; Dementia; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction | interventions — Positron-Emission Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: PET Scan
  Other Names: Collection of institutional practice PET imaging data

SUMMARY:
The Imaging Dementia-Evidence for Amyloid Scanning (IDEAS) Study will establish an open-label, longitudinal cohort study to assess the impact of amyloid PET on patient outcomes. The study will be performed in accordance with the Center for Medicare & Medicaid Services (CMS) policy of Coverage with Evidence Development (CED) in Medicare beneficiaries who meet the Appropriate Use Criteria (AUC) for amyloid PET (Johnson et al. 2013). Our hypothesis is that amyloid PET will decrease uncertainty and increase confidence in the underlying cause of cognitive impairment, that this will translate into earlier counseling and interventions in these domains, and that these interventions will lead to improved outcomes.

DETAILED DESCRIPTION:
The IDEAS Study is an observational, open-label, longitudinal cohort study designed to assess the impact of amyloid PET on patient-oriented outcomes in Medicare beneficiaries with mild cognitive impairment (MCI) or dementia of uncertain etiology. The study falls under the Centers for Medicare & Medicaid Services (CMS) Coverage with Evidence Development (CED) policy. A total of 18,488 Medicare beneficiaries meeting Appropriate Use Criteria (AUC) for amyloid PET will be enrolled over 24 months at sites throughout the United States. Dementia specialists will team with PET facilities able to perform amyloid PET and with trained radiologists/nuclear medicine physicians, all of whom will consent to completing the data requirements and timelines for the study. Amyloid PET will be performed and interpreted at each facility with results provided to the ordering physician for support in further clinical decision making, which will be captured for the study.

Our over-arching hypothesis is that, in diagnostically uncertain cases, knowledge of amyloid status as determined by amyloid PET will lead to significant changes in patient management, and that this will translate into improved long-term outcomes. We will pursue two specific aims:

Aim 1 investigates the impact of amyloid PET on short-term patient management, by comparing pre-PET intended management (ascertained in a case report form [CRF] prior to PET) to post-PET actual management 90-days post-PET). The primary objective will be to test whether amyloid PET leads to a ≥ 30% change between intended and actual patient management within 90 days in a cumulative endpoint consisting of: Alzheimer's disease (AD) drug therapy, other drug therapy, and counseling about safety and future planning. Secondary objectives will assess the impact of amyloid PET results on clinical diagnosis and prevention of unnecessary diagnostic procedures and treatments.

Aim 2 utilizes Medicare claims data to compare medical outcomes at 12 months for patients enrolled in the longitudinal cohort (amyloid PET-known) with those for a matched control cohort of patients who have never undergone amyloid PET imaging (amyloid PET-naïve). The primary objective will be to determine if amyloid PET in the amyloid PET-known cohort of patients is associated with a ≥ 10% reduction in hospitalizations and emergency room visits in comparison to the matched amyloid PET-naïve patients. Secondary objectives will examine whether knowledge of amyloid PET status reduces hospitalizations related to ambulatory-sensitive conditions, whether the association between amyloid PET knowledge and health outcomes varies by baseline cognitive status (MCI versus dementia) and amyloid status (amyloid positive versus negative). The amyloid PET-naïve cohort will be identified via a matching algorithm where each individual in the amyloid PET-known cohort will be matched to one individual with similar dementia diagnosis, pre-scan dementia-related resource utilization, age, race, gender, ethnicity, geographic location, and comorbid chronic conditions likely to impact cognition or the outcomes of interest seen at the same time as the amyloid PET-known patient (concurrent control).

In pursuing these Aims, we will generate valuable observational data on clinical utility that will inform future use of this technology in diagnostic algorithms, and develop a cohort of patients who undergo amyloid PET and can serve as a foundation to address future research questions.

ELIGIBILITY:
Inclusion Criteria:

* 65 and older;
* Medicare beneficiary;
* Diagnosis of MCI or dementia, according to DSM-IV and/or National Institutes of Aging-Alzheimer's Association criteria, verified by a dementia specialist within 24 months (American Psychiatric Association. 2000; McKhann et al. 2011; Albert et al. 2011);
* Meets AUC:
* Cognitive complaint verified by objectively confirmed cognitive impairment;
* The etiologic cause of cognitive impairment is uncertain after a comprehensive evaluation by a dementia specialist, including general medical and neurological examination, mental status testing including standard measures of cognitive impairment, laboratory testing, and structural neuroimaging as below;
* Alzheimer's disease is a diagnostic consideration;
* Knowledge of amyloid PET status is expected to alter diagnosis and management.
* Head MRI and/or CT within 24 months prior to enrollment;
* Clinical laboratory assessment (complete blood count [CBC], standard blood chemistry profile, thyroid stimulating hormone [TSH], vitamin B12) within the 12 months prior to enrollment;
* Able to tolerate amyloid PET required by protocol, to be performed at a participating PET facility;
* English or Spanish speaking (for the purposes of informed consent);
* Willing and able to provide consent. Consent may be by proxy.

Exclusion Criteria:

* Normal cognition or subjective complaints that are not verified by cognitive testing.
* Knowledge of amyloid status, in the opinion of the referring dementia expert, may cause significant psychological harm or otherwise negatively impact the patient or family.
* Scan is being ordered solely based on a family history of dementia, presence of apolipoprotein E, or in lieu of genotyping for suspected autosomal mutation carriers.
* Scan being ordered for nonmedical purposes (e.g., legal, insurance coverage, or employment screening).
* Cancer requiring active therapy (excluding non-melanoma skin cancer);
* Hip/pelvic fracture within the 12 months prior to enrollment;
* Body weight exceeds PET scanner weight limit;
* Life expectancy less than 24 months based on medical co-morbidities;
* Residence in a skilled nursing facility.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Participants must be Medicare beneficiaries referred by qualified dementia specialists and must meet AUC for amyloid PET (Johnson et al. 2013).
Sampling Method: Non-Probability Sample
Enrollment: 18488 (Actual)
Dates: Start 2016-02; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
To assess the impact of amyloid PET on the management of patients meeting Appropriate Use Criteria (AUC) | 90 days
  Test whether amyloid PET imaging will lead to a ≥ 30% change between intended and actual patient management within 90 days in a composite measure of at least one of the following:
  1. AD drug therapy;
  2. Other drug therapy; and
  3. Counseling about safety and future planning.
To assess the impact of amyloid PET on hospital admissions and emergency room visits in patients enrolled in the cohort (amyloid PET-known) compared to matched patients not in the cohort (amyloid PET-naïve) over 12 months | 12 months
  Determine if amyloid PET is associated with a ≥ 10% relative reduction in amyloid PET-known patients in comparison to matched amyloid PET-naïve patients in the following:
  1. Inpatient hospital admissions over 12 months.
  2. Emergency room visits over 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Gil D Rabinovici, MD, Study Chair — University of California, San Francisco
Locations (2):
- United States (2):
  - American College of Radiology Imaging Network, Philadelphia, Pennsylvania
  - Https://Www.Ideas-Study.Org/Site-Locator/, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Johnson KA, Minoshima S, Bohnen NI, Donohoe KJ, Foster NL, Herscovitch P, Karlawish JH, Rowe CC, Hedrick S, Pappas V, Carrillo MC, Hartley DM. Update on appropriate use criteria for amyloid PET imaging: dementia experts, mild cognitive impairment, and education. J Nucl Med. 2013 Jul;54(7):1011-3. doi: 10.2967/jnumed.113.127068. Epub 2013 Jun 10. PMID 23753186
- [Background] Thies W and Bleiler L. (2013).
- [Background] Naylor MD, Karlawish JH, Arnold SE, et al. (2012).
- [Background] Phelan EA, Borson S, Grothaus L, Balch S, Larson EB. Association of incident dementia with hospitalizations. JAMA. 2012 Jan 11;307(2):165-72. doi: 10.1001/jama.2011.1964. PMID 22235087
- [Background] Feng Z, Coots LA, Kaganova Y, Wiener JM. Hospital and ED use among Medicare beneficiaries with dementia varies by setting and proximity to death. Health Aff (Millwood). 2014 Apr;33(4):683-90. doi: 10.1377/hlthaff.2013.1179. PMID 24711331
- [Background] Fisher GG, Franks MM, Plassman BL, Brown SL, Potter GG, Llewellyn D, Rogers MA, Langa KM. Caring for individuals with dementia and cognitive impairment, not dementia: findings from the aging, demographics, and memory study. J Am Geriatr Soc. 2011 Mar;59(3):488-94. doi: 10.1111/j.1532-5415.2010.03304.x. PMID 21391939
- [Background] Clark DO, Stump TE, Tu W, Miller DK, Langa KM, Unverzagt FW, Callahan CM. Hospital and nursing home use from 2002 to 2008 among U.S. older adults with cognitive impairment, not dementia in 2002. Alzheimer Dis Assoc Disord. 2013 Oct-Dec;27(4):372-8. doi: 10.1097/WAD.0b013e318276994e. PMID 23151595
- [Background] Schaller S, Mauskopf J, Kriza C, Wahlster P, Kolominsky-Rabas PL. The main cost drivers in dementia: a systematic review. Int J Geriatr Psychiatry. 2015 Feb;30(2):111-29. doi: 10.1002/gps.4198. Epub 2014 Oct 16. PMID 25320002
- [Background] Hurd MD, Martorell P, Delavande A, Mullen KJ, Langa KM. Monetary costs of dementia in the United States. N Engl J Med. 2013 Apr 4;368(14):1326-34. doi: 10.1056/NEJMsa1204629. PMID 23550670
- [Background] Connell CM, Gallant MP. Spouse caregivers' attitudes toward obtaining a diagnosis of a dementing illness. J Am Geriatr Soc. 1996 Aug;44(8):1003-9. doi: 10.1111/j.1532-5415.1996.tb01881.x. PMID 8708288
- [Background] Klein E and Karlawish J. (2013).
- [Background] Elson P. Do older adults presenting with memory complaints wish to be told if later diagnosed with Alzheimer's disease? Int J Geriatr Psychiatry. 2006 May;21(5):419-25. doi: 10.1002/gps.1485. PMID 16676286
- [Background] Carpenter BD, Xiong C, Porensky EK, Lee MM, Brown PJ, Coats M, Johnson D, Morris JC. Reaction to a dementia diagnosis in individuals with Alzheimer's disease and mild cognitive impairment. J Am Geriatr Soc. 2008 Mar;56(3):405-12. doi: 10.1111/j.1532-5415.2007.01600.x. Epub 2008 Jan 5. PMID 18194228
- [Background] Knopman DS, DeKosky ST, Cummings JL, Chui H, Corey-Bloom J, Relkin N, Small GW, Miller B, Stevens JC. Practice parameter: diagnosis of dementia (an evidence-based review). Report of the Quality Standards Subcommittee of the American Academy of Neurology. Neurology. 2001 May 8;56(9):1143-53. doi: 10.1212/wnl.56.9.1143. PMID 11342678
- [Background] American Psychiatric Association. Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR). 2000.
- [Background] McKhann GM, Knopman DS, Chertkow H, Hyman BT, Jack CR Jr, Kawas CH, Klunk WE, Koroshetz WJ, Manly JJ, Mayeux R, Mohs RC, Morris JC, Rossor MN, Scheltens P, Carrillo MC, Thies B, Weintraub S, Phelps CH. The diagnosis of dementia due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):263-9. doi: 10.1016/j.jalz.2011.03.005. Epub 2011 Apr 21. PMID 21514250
- [Background] Albert MS, DeKosky ST, Dickson D, Dubois B, Feldman HH, Fox NC, Gamst A, Holtzman DM, Jagust WJ, Petersen RC, Snyder PJ, Carrillo MC, Thies B, Phelps CH. The diagnosis of mild cognitive impairment due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):270-9. doi: 10.1016/j.jalz.2011.03.008. Epub 2011 Apr 21. PMID 21514249
- [Background] Bradford A, Kunik ME, Schulz P, Williams SP, Singh H. Missed and delayed diagnosis of dementia in primary care: prevalence and contributing factors. Alzheimer Dis Assoc Disord. 2009 Oct-Dec;23(4):306-14. doi: 10.1097/WAD.0b013e3181a6bebc. PMID 19568149
- [Background] Beach TG, Monsell SE, Phillips LE, Kukull W. Accuracy of the clinical diagnosis of Alzheimer disease at National Institute on Aging Alzheimer Disease Centers, 2005-2010. J Neuropathol Exp Neurol. 2012 Apr;71(4):266-73. doi: 10.1097/NEN.0b013e31824b211b. PMID 22437338
- [Background] Zilkens RR, Duke J, Horner B, Semmens JB, Bruce DG. (2014).
- [Background] Bei Hu, Ross L, Neuhaus J, Knopman D, Kramer J, Boeve B, Caselli RJ, Graff-Radford N, Mendez MF, Miller BL, Boxer AL. Off-label medication use in frontotemporal dementia. Am J Alzheimers Dis Other Demen. 2010 Mar;25(2):128-33. doi: 10.1177/1533317509356692. Epub 2010 Feb 1. PMID 20124256
- [Background] Mendez MF, Shapira JS, McMurtray A, Licht E. Preliminary findings: behavioral worsening on donepezil in patients with frontotemporal dementia. Am J Geriatr Psychiatry. 2007 Jan;15(1):84-7. doi: 10.1097/01.JGP.0000231744.69631.33. PMID 17194818
- [Background] Boxer AL, Knopman DS, Kaufer DI, et al. (2013).
- [Background] Doody RS, Thomas RG, Farlow M, et al. Alzheimer's Disease Cooperative Study Steering and G. Solanezumab Study (2014).
- [Background] Salloway S, Sperling R, Fox NC, et al. (2014).
- [Background] Kirson NY, Hunter CA, Desai U, et al. (2013). "Excess costs associated with a misdiagnosis of Alzheimer's disease among U.S. Medicare beneficiaries with vascular dementia or Parkinson's disease." Alzheimer's Association International Conference. Boston, MA.
- [Background] Geldmacher DS, Kirson NY, Birnbaum HG, et al. (2014).
- [Background] Johnson KA, Minoshima S, Bohnen NI, et al. (2013).
- [Background] Frederiksen KS, Hasselbalch SG, Hejl AM, Law I, Hojgaard L, Waldemar G. Added Diagnostic Value of (11)C-PiB-PET in Memory Clinic Patients with Uncertain Diagnosis. Dement Geriatr Cogn Dis Extra. 2012 Jan;2(1):610-21. doi: 10.1159/000345783. Epub 2012 Dec 13. PMID 23341826
- [Background] Ossenkoppele R, Prins ND, Pijnenburg YA, et al. (2013).
- [Background] Grundman M, Pontecorvo MJ, Salloway SP, et al. (2013).
- [Background] Sanchez-Juan P, Ghosh PM, Hagen J, et al. (2014).
- [Background] Bynum JP, Rabins PV, Weller W, Niefeld M, Anderson GF, Wu AW. The relationship between a dementia diagnosis, chronic illness, medicare expenditures, and hospital use. J Am Geriatr Soc. 2004 Feb;52(2):187-94. doi: 10.1111/j.1532-5415.2004.52054.x. PMID 14728626
- [Background] Schwarzkopf L, Menn P, Leidl R, et al. (2012).
- [Background] Toot S, Devine M, Akporobaro A, Orrell M. Causes of hospital admission for people with dementia: a systematic review and meta-analysis. J Am Med Dir Assoc. 2013 Jul;14(7):463-70. doi: 10.1016/j.jamda.2013.01.011. Epub 2013 Mar 17. PMID 23510826
- [Background] Lyketsos CG, Sheppard JM, Rabins PV. Dementia in elderly persons in a general hospital. Am J Psychiatry. 2000 May;157(5):704-7. doi: 10.1176/appi.ajp.157.5.704. PMID 10784461
- [Background] Shen HN, Lu CL, Li CY. (2012).
- [Background] Lyketsos CG. Prevention of unnecessary hospitalization for patients with dementia: the role of ambulatory care. JAMA. 2012 Jan 11;307(2):197-8. doi: 10.1001/jama.2011.2005. No abstract available. PMID 22235092
- [Derived] Rabinovici GD, Gatsonis C, Apgar C, Chaudhary K, Gareen I, Hanna L, Hendrix J, Hillner BE, Olson C, Lesman-Segev OH, Romanoff J, Siegel BA, Whitmer RA, Carrillo MC. Association of Amyloid Positron Emission Tomography With Subsequent Change in Clinical Management Among Medicare Beneficiaries With Mild Cognitive Impairment or Dementia. JAMA. 2019 Apr 2;321(13):1286-1294. doi: 10.1001/jama.2019.2000. PMID 30938796